CLINICAL TRIAL: NCT04067531
Title: Treatment of BV With First Deqularum and Then Direkt After With Vaginal Clindamycin Cream.
Brief Title: Treatment of BV With First Deqularum and Then Direkt After Clindamycin
Acronym: BV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, professor, Skaraborg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-03

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment of BV (Other): all patients be treated with first Deqularum then with clindamycin Cream,
  Interventions: Drug: treatment of BV with first Deqularum and then direkt after with vaginal clindamycin

INTERVENTIONS:
Drug: treatment of BV with first Deqularum and then direkt after with vaginal clindamycin — All patients will get the same treatment

SUMMARY:
Treatment of BV with first deqularum cloride and then followed with clindamycin vaginal Cream.

DETAILED DESCRIPTION:
The hypoteses is that deqularum cloride takes away the biofilm so that clindamycin will kills the bacteria.

Cure rate will be followed up after 1 month and then after 6 month

ELIGIBILITY:
Inclusion Criteria:

* healthy women with BV

Exclusion Criteria:

* women treated with antibiotics within 1 month

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
cure of BV | 6 month
  cure rate of BV

CONTACTS AND LOCATIONS:
Overall Officials: P-G Larsson, Principal Investigator — professor
Locations (1):
- Department of Ob/Gyn, Skaraborgshospital Skövde, Skövde, Sweden